CLINICAL TRIAL: NCT04370522
Title: The NIKOLE Study: Characterization of Innate Immune System in Patients With Luminal Advanced Breast Cancer
Brief Title: Characterization of Innate Immune System in Patients With Luminal Advanced Breast Cancer
Acronym: NIKOLE
Status: Active, not recruiting | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2018-03
Record Dates: First submitted 2020-04-24; First posted 2020-05-01 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Luminal; HER2 negative; Endocrine therapy resistance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Plasma, Peripheral Blood Mononuclear Cells and tumor tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: hormone-sensitive disease: Patients who initiate ET in first line of advanced disease, they could be patients de novo with no previous ET or patients who received adjuvant ET and experience disease recurrence more than one year after its completion.
  Patients will be divided in two subgroups according to having or not received previous ET.
- Cohort B: hormone-resistant disease: Patients in progression who are starting a first or second line of ET for advanced Breast Cancer (BC) and showing one of following the hormone-resistance criteria to any ET:
  For first line:
  * Primary hormone-resistance: disease recurrence occurs within the first two years of adjuvant ET.
  * Secondary hormone-resistance: disease recurrence occurs after the first two years of adjuvant ET or during the first year after its completion.
  For second line:
  * Primary hormone-resistance: disease progression occurs within the first 6 months of ET for advanced disease.
  * Secondary hormone-resistance: disease progression occurs after the first 6 months of ET for advanced disease.
  Patients will be divided in two subgroups according to having primary or secondary hormone-resistance.

SUMMARY:
This is a multicentre, prospective, observational, no post-authorization study. This study will be opened for recruitment approximately for 12 months for a pilot phase including at least 25-30 patients and 6 controls and for 12 additional months to complete patient and control inclusion until 90 patients and 20 control depending on the first part study results.

DETAILED DESCRIPTION:
After enrolment, patients will be assigned to one of the following cohorts according to their level of hormone-resistance:

* Cohort A (hormone-sensitive disease).
* Cohort B (hormone-resistant disease).

In both cohorts it will be collected residual pre-treatment tumor samples from metastatic lesions, preferably obtained after last treatment just prior to study entry, and/or primary breast tumor; as well as serial blood samples at baseline, after 6 weeks, at the same time of radiological re-evaluation (3 months after ET initiation) and at progressive disease (PD) which will be used for serial analytic determinations of the expression profiles of Natural Killer (NK) cells, other lymphoid innate cells, NKG2D ligands, cytokines and other possible biomarkers; in addition to obtain local data of hemogram and estradiol, Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) levels.

Patients who have participated in the study during their first line of ET are eligible to participate after progression, when they initiate the second line of ET (in this case, inclusion/exclusion criteria should be checked newly and Informed Consent Form (ICF) signed again).

From the control population it will be collected blood and local data (e.g. hemogram, estradiol, FSH and LH levels), in a single time-point after ICF signature.

ELIGIBILITY:
INCLUSION AND EXCLUSION CRITERIA OF PATIENTS

Inclusion Criteria:

1. Female ≥ 18 years of age on day of signing informed consent.
2. Patient with histological confirmation of BC with evidence of metastatic or advanced disease not amenable to resection or radiation therapy with curative intent.
3. Documented Hormonal Receptor (HR) positive status based on local testing (preferably assessed on the most recent tumour biopsy available). HR+ is defined as ≥ 1% positive cells by immuno-histochemistry (IHC) for ER and/or Progesterone Receptor (PgR).
4. Documented HER2 negative status based on local testing (preferably assessed on the most recent tumour biopsy available). HER2- is defined as IHC score 0/1+ or negative by in situ hybridization according to local criteria.
5. Patients who are going to receive ET in first or second line for advanced disease (in monotherapy or in combination). It is allowed the inclusion of patients that have received or are going to initiate tamoxifen, Luteinizing Hormone Releasing Hormone (LHRH) analogues, aromatase inhibitors or fulvestrant. It is also possible to recruit patients that have received or are going to initiate cyclin or mTOR inhibitors in combination with ET. (NOTE: it is not allowed the inclusion of patients after first line of chemotherapy that are in response and initiate maintenance ET).
6. Patients who have participated in the study during their first line of ET are eligible to participate again when they receive the second line of ET (in this case eligibility criteria should be checked newly and ICF signed again).
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
8. Patient must have a life expectancy ≥ 16 weeks.
9. The patient has signed and dated the ICF for study participation.
10. Willingness and ability to comply with the protocol for the duration of the study including biological sample collection.

Exclusion Criteria:

1. Have received more than 1 prior therapy line for advanced BC disease.
2. Have received chemotherapy with response and initiate ET as maintenance treatment.
3. Locally advanced breast cancer.
4. Previous or concomitant treatment with immunotherapeutic agents.
5. Major surgical procedure unrelated to breast cancer or significant traumatic injury within 28 days prior to study entry.
6. History of concurrent or previously treated non-breast malignancies except for appropriately treated 1) non-melanoma skin cancer and/or 2) in situ carcinomas, including cervix and colon.
7. Has a diagnosis of immunodeficiency, autoimmune disease or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of ET.
8. Has an active infection requiring systemic therapy. Patients with solved infection that has finished antibiotic treatment within 7 days prior to study entry could be included.
9. Has a known history of active Tuberculosis Bacillus (TB) or Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or a known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (HCV) (e.g. HCV RNA [qualitative] is detected).
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
11. There is evidence that the patient is pregnant or breastfeeding, or patient is expecting to conceive within the projected duration of the study.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the investigator.

In the case of values of Neutrophil Count (NC) < 1.5 x 109/L prior to study entry or in case of patients who have received or are going to receive an investigational product, the information about NC or the investigational product should be checked with chief investigator in order to check any possible interference with the study results.

INCLUSION CRITERIA OF CONTROL PARTICIPANTS

1. Female ≥ 18 years of age on day of signing informed consent.
2. The participant has signed and dated the ICF for study participation.
3. Absence of evidences of current tumor malignancies or active infectious disease.
4. Absence of history or current evidences of immunological and rheumatologic diseases or any condition, therapy, or laboratory abnormality that might confound the results of the study, in the opinion of the investigator.
5. Willingness and ability to comply with blood and study data collection.
6. To have data to be able to be classified as pre- o postmenopausal.

Postmenopausal women are defined as women fulfilling any one of the following criteria (based on the National Comprehensive Cancer Network (NCCN) definition of menopause [NCCN 2008]):

* Prior bilateral oophorectomy.
* Age > 60 years.
* Age ≤ 60 years and with amenorrhea for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and FSH and estradiol in the postmenopausal range.

Women who didn't comply with any of the prior criteria will be considered premenopausal women for the purposes of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Luminal/HER2 negative advanced Breast Cancer patients and a control group of healthy women (premenopausal and postmenopausal).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Amount of innate immune cells | Up to disease progression, an average of 25 months
  Amount of the different populations of innate immune cells (e.g. NK cells, ILC1, ILC2 and ILC3) detected in tumor tissue and/or serial peripheral blood samples.
  Blood samples will be collected from the patients at the following time-points: at baseline, after 6 weeks, at tumor re-evaluation of treatment and after end of therapy (before the beginning of the next treatment).
  Blood samples will be collected from the control participants in a single time-point after signature of the corresponding Inform Consent Form.
  It is required the shipment of residual pre-treatment tumor samples (leftover from medical routine assistance) from primary and/or the recurrence/metastatic sites, preferably obtained after the last treatment prior to study entry.
Activation level of innate immune cells | Up to disease progression, an average of 25 months
  Activation level of the different populations of innate immune cells (e.g. NK cells, ILC1, ILC2 and ILC3) detected in tumor tissue and/or serial peripheral blood samples.
  Blood samples will be collected from the patients at the following time-points: at baseline, after 6 weeks, at tumor re-evaluation of treatment and after end of therapy (before the beginning of the next treatment).
  Blood samples will be collected from the control participants in a single time-point after signature of the corresponding Inform Consent Form.
  It is required the shipment of residual pre-treatment tumor samples (leftover from medical routine assistance) from primary and/or the recurrence/metastatic sites, preferably obtained after the last treatment prior to study entry.
Analyses of the expression level of cytokines and/or rNKG2D ligands | Up to disease progression, an average of 25 months
  Analyses of the expression level of cytokines and/or rNKG2D ligands in tumor tissue and/or serial peripheral blood samples.
  Blood samples will be collected from the patients at the following time-points: at baseline, after 6 weeks, at tumor re-evaluation of treatment and after end of therapy (before the beginning of the next treatment).
  Blood samples will be collected from the control participants in a single time-point after signature of the corresponding Inform Consent Form.
  It is required the shipment of residual pre-treatment tumor samples (leftover from medical routine assistance) from primary and/or the recurrence/metastatic sites, preferably obtained after the last treatment prior to study entry.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in relation with values of innate immune cells, cytokines and ligands of rNKG2D | Up to disease progression, an average of 25 months
  Progression Free Survival (PFS) defined as the time from the start of therapy to the first documented progressive disease, or death from any cause, whichever occurs first. Progressive disease will be based on the investigator's assessment according to the standard institutional guidelines, and following as much as possible RECIST version 1.1. Tumor assessment during treatment will be performed according the clinical standard of care and following as much as possible RECIST version 1.1. every 3 months (+/- 1 month).
Objective Response Rate (ORR) in relation with values of innate immune cells, cytokines and ligands of rNKG2D | Up to disease progression, an average of 25 months
  OR rate (ORR) is defined as the Complete Response (CR) + Partial Response (PR) out of the patients who had measurable disease at baseline, according to the standard institutional guidelines and following as much as possible the RECIST version 1.1. Tumor assessment during treatment will be performed according the clinical standard of care and following as much as possible RECIST version 1.1. every 3 months (+/- 1 month).
Clinical Benefit (CB) in relation with values of innate immune cells, cytokines and ligands of rNKG2D | Up to disease progression, an average of 25 months
  Clinical Benefit (CB): is defined as complete response (CR), partial response (PR), or stable disease (SD) lasting more than 24 weeks; based on the investigator's assessment according to the standard institutional guidelines, and following as much as possible according to the RECIST version 1.1. The definition of Response/non-Response and Stable Disease will be based on the RECIST version 1.1. Tumor assessment during treatment will be performed according the clinical standard of care and following as much as possible RECIST version 1.1. every 3 months (+/- 1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Morales Meseguer
Locations (2):
- Spain (2):
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- See also: GEICAM is the Spanish Breast Cancer Research Group — http://www.geicam.org